CLINICAL TRIAL: NCT03894475
Title: Non-inferiority of Portable Versus Desktop Spirometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Collaborators: Healthup Sp. z o.o. (Industry)
Responsible Party: Principal Investigator, Piotr Boros, Prof. Piotr Boros, M.D., Ph.D., National Institute for Tuberculosis and Lung Diseases, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KB-6
Record Dates: First submitted 2019-03-19; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Asthma; COPD
Keywords: Asthma; COPD; Mobile Spirometry
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Active Comparator): Patient would first perform an examination with handheld spirometer (AioCare), followed by measurements with the reference spirometer (MGC)
  Interventions: Device: AioCare; Device: Spirometer USB CPFS/D (MGC Diagnostics)
- Sequence B (Active Comparator): Patient would first perform an examination with the reference spirometer (MGC), followed by measurements with handheld spirometer (AioCare)
  Interventions: Device: AioCare; Device: Spirometer USB CPFS/D (MGC Diagnostics)

INTERVENTIONS:
Device: AioCare — AioCare is an ultraportable, handheld hardware module that contains the MEMS-based flow sensor and electronics, with a dedicated mobile application that works on iOS and Android operating systems. The unit is used with a disposable mouthpiece fitted to the tip of the flow tube, and a nose clip. AioCare is connected to its dedicated mobile application, which contains software that will show flow-volume graphs and results in real time. The device encompasses all of the widely used spirometry parameters, including: peak expiratory flow (PEF), forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), FEV1/FVC ratio, forced expiratory flow at 25% of expiration (FEF25), forced expiratory flow at 50% of expiration (FEF50), forced expiratory flow at 75% of expiration (FEF75), and forced expiratory volume in 6 second (FEV6).
Device: Spirometer USB CPFS/D (MGC Diagnostics) — Spirometer USB CPFS/D (MGC Diagnostics) is a diagnostic desktop spirometer used in hospitals/clinics. CPFS/D USB spirometer is compatible with desktop and laptop computers.

SUMMARY:
The investigators compared the ventilation parameters for volume and flow obtained from standard spirometry procedures from patients presently monitored and treated for asthma or chronic obstructive pulmonary disease (COPD) using AioCare (HealthUp Sp. z o.o., Serial Number: MS082017005412, software version: MySpiroo app 1.1.14) as the tested device and Spirometer USB CPFS/D (MGC Diagnostics) as the reference, which required calibration prior to each session. Spirometry measurements were performed on sixty-two patients (forty-four females (58±17 years old) and eighteen males (52±19 years old)) at the Institute of Tuberculosis and Lung Disease in Warsaw, Poland. Participants were asked to perform correct spirometry examinations (which means at least three technically correct exhales and meeting repeatability criteria for FEV1 and FVC) on both measuring devices with a five-minute break between devices to prevent respiratory muscle fatigue. The highest value from all acceptable spirometry results was then used for analysis. All spirometry examinations followed ERS/ATS standards.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18.
2. Diagnosed asthma or COPD
3. Signed consent to participation in the research experiment.
4. Ability to comply with the spirometry protocol.

Exclusion Criteria:

1. Pregnant females (based on declaration; no pregnancy tests are planned before the test).
2. Recent myocardial infarction (<30 days).
3. Known thoracic, aortic or cerebral aneurysm.
4. Recent stroke, eye surgery, thoracic/abdominal surgery.
5. Haemoptysis.
6. Recent pneumothorax.
7. Uncontrolled hypertension.
8. Pulmonary Embolism.
9. Angina.
10. Chest or abdominal pain of any etiology.
11. Oral or facial pain exacerbated by a mouthpiece.
12. Stress incontinence.
13. Dementia or state of confusion. 14, Acute Diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of PEF between AioCare and CPFS/D USB Spirometer | 6 months
  Comparison of Peak Expiratory Flow obtained during a standard dynamic spirometry measured with AioCare (HealthUp) and reference spirometer (MGC)
Non-inferiority of FEV1 between AioCare and CPFS/D USB Spirometer | 6 months
  Comparison of Forced Expiratory Volume in the first second (FEV1) obtained during a standard dynamic spirometry measured with AioCare (HealthUp) and reference spirometer (MGC)
Non-inferiority of FVC between AioCare and CPFS/D USB Spirometer | 6 months
  Comparison of Forced Vital Capacity (FVC) obtained during a standard dynamic spirometry measured with AioCare (HealthUp) and reference spirometer (MGC)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Boros, Prof. dr hab. n. med., Principal Investigator — National Institute for Tuberculosis and Lung Diseases, Poland
Locations (1):
- National Institute for Tuberculosis and Lung Diseases, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided